CLINICAL TRIAL: NCT06697158
Title: Investigation of the Effects of Complex Decongestive Physiotherapy on Sleep Quality and Quality of Life in Women With Breast Cancer Related Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif Duygu, PT PhD, Abant Izzet Baysal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAIBU-FTR-ED-003
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: Breast Cancer-Related Lymphedema; Physiotherapy and Rehabilitation; Sleep Quality; Local Tissue Fluid; Quality of Life
MeSH Terms: conditions — Breast Cancer Lymphedema; Sleep Initiation and Maintenance Disorders | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): This study is planned as a prospective quasi-experimental design (pre-test, intervention, post-test). The study will be conducted at the Women's Health and Lymphedema Unit of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Abant İzzet Baysal University, Bolu, Turkey. All participants will provide written informed consent before participating in the study.
  Participants The study aims to include a total of 31 patients who develop unilateral upper extremity lymphedema following breast cancer surgery. The inclusion criterion for lymphedema diagnosis will be a difference of more than 2 cm in circumferential measurements between both arms. Only individuals diagnosed with lymphedema by a physician will be included in the study.
  Interventions: Other: Physiotherapy and rehabilitation

INTERVENTIONS:
Other: Physiotherapy and rehabilitation — Complex Decongestive Physiotherapy (CDP) Complex Decongestive Physiotherapy (CDP) consists of Manual Lymphatic Drainage (MLD), skin care, compression bandaging, and exercise, which are routinely used in clinical practice (9). CDP sessions will last approximately one hour each and will be administered for 4 weeks, with 5 sessions per week, totaling 20 sessions.
  Manual Lymphatic Drainage (MLD) is a massage technique involving rhythmic, gentle pressure movements aimed at reducing the accumulation of lymphatic fluid in conditions such as lymphedema. This therapy facilitates the drainage of lymphatic fluid into the body's primary lymphatic pathways, thereby reducing edema, pain, and tightness, while enhancing range of motion and overall quality of life. MLD typically focuses on areas with a high concentration of lymph nodes, promoting the smooth circulation of lymph fluid. Treatment sessions usually last between 30 minutes to one hour.
  Other Names: Complex Decongestive Physiotherapy

SUMMARY:
Breast cancer is the most common type of cancer among women globally and has the highest mortality rate. Surgical interventions are typically required in the treatment of breast cancer, but these procedures can lead to complications such as infection, seroma, hematoma, cellulitis, and particularly lymphedema due to disruptions in the physiology of axillary lymphatic vessels.

Breast Cancer-Related Lymphedema (BCRL) commonly develops within the first two years following surgical intervention and its incidence varies depending on the surgical method used. The incidence of lymphedema after Sentinel Lymph Node Biopsy (SLNB) is around 5%, whereas it increases to 30-50% after Axillary Lymph Node Dissection (ALND).

BCRL significantly impacts the quality of life (QoL) through physical symptoms such as swelling, pain, tightness, and limited range of motion, as well as psychosocial issues including depression, social isolation, and sleep disturbances. Sleep disorders, in particular, are associated with depression and contribute to a further decline in QoL.

In the treatment of BCRL, both conservative (non-surgical) and surgical methods are traditionally employed. Complex Decongestive Physiotherapy (CDP) is considered the gold standard for the conservative management of lymphedema. CDP comprises a two-phase treatment process. The first phase, known as the "Decongestion Phase," generally lasts 2-4 weeks and includes manual lymphatic drainage (MLD), skin care, compression therapy with multi-layered short-stretch bandages, and muscle-pumping exercises. The second phase, the "Maintenance Phase," is more prolonged and aims to sustain the results achieved in Phase 1. It includes compression with low-stretch elastic garments, skin care, exercises, and patient-administered MLD as needed.

The primary objectives of CDP are to improve lymphatic circulation, reduce swelling, pain, and tightness, increase the range of motion, and ultimately improve the QoL. Studies have shown that CDP significantly enhances sleep quality and QoL in women with BCRL.

However, most existing studies examine all stages of BCRL without comparing the effects of CDP across different stages. The impact of CDP on sleep and QoL may vary depending on the stage of BCRL, highlighting the need for specific research on its effects in particular populations. Furthermore, many studies lack follow-up data, leaving the Maintenance Phase of CDP largely unexplored.

This study aims to investigate the effects of CDP, including both the Decongestion and Maintenance phases, on sleep quality and QoL specifically in women with Stage II BCRL.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer and has the highest mortality rate among women worldwide. According to the 2022 Global Cancer Observatory statistics, breast cancer affects approximately 20 million women globally. It accounts for 23.8% of all cancers in women, making it the most frequently diagnosed type (1). Various treatment options are available for breast cancer patients. Most breast cancer cases require surgical procedures for advanced diagnosis and treatment. However, these procedures may lead to complications such as infection, seroma, hematoma, cellulitis, and, most importantly, lymphedema due to disruption in the physiology of axillary lymphatic vessels (2).

Lymphedema is a chronic disease characterized by the accumulation of lymphatic fluid, leading to skin and tissue changes. It results from lymphatic system insufficiency and impaired lymph transport (3, 4). Lymphedema occurs due to the buildup of excess water, filtered plasma proteins, extravascular blood cells, and products of parenchymal and stromal cells in the extracellular space (3).

Breast Cancer-Related Lymphedema (BCRL) often develops within two years following breast cancer diagnosis or surgery (5). The incidence of BCRL varies depending on the surgical method used for diagnosis and treatment. While the rate of lymphedema following Sentinel Lymph Node Biopsy (SLNB) is around 5%, it increases to 30-50% after Axillary Lymph Node Dissection (ALND). When ALND is combined with Regional Node Irradiation (RNI), the rate reaches 20-50% (2). One study identified ALND as the primary trigger for BCRL and emphasized avoiding this procedure whenever possible (6). Risk factors for BCRL include ALND, radiotherapy (RT), chemotherapy, postoperative seroma, obesity/high body mass index, smoking, total mastectomy, and postoperative bleeding (7, 8).

Clinically, BCRL manifests as chronic swelling, localized pain, heaviness, and tightness (9). It significantly impacts the quality of life (QoL) and causes psychosocial issues such as depression, social isolation, and decreased sleep quality in addition to physical symptoms like swelling, heaviness, tightness, and reduced range of motion (7). Pain in the affected limb makes it difficult for patients to fall asleep. Overuse of the dominant limb can exacerbate symptoms like swelling, pain, heaviness, stiffness, and numbness, further disrupting sleep quality. Sleep disturbances in BCRL patients are associated with depression and lower QoL scores. A study by Tamam et al. also reported a significant decline in both QoL and sleep quality among women with varying stages of BCRL (10, 11).

The treatment of BCRL is traditionally divided into conservative (non-operative) and operative methods (3). Complex Decongestive Physiotherapy (CDP) is considered the gold standard for conservative treatment of lymphedema. This non-invasive approach consists of two phases. Phase 1, known as the "Decongestion Phase", includes skin care, manual lymphatic drainage (MLD), compression therapy with multi-layered short-stretch bandages, and muscle-pumping exercises. Phase 2, the "Maintenance Phase", aims to preserve and optimize the results achieved in Phase 1. It involves compression with a low-stretch elastic garment, skin care, exercises, and patient-administered MLD as needed. Phase 1 typically lasts 2-4 weeks, while Phase 2 can extend for months or even years (3, 12, 13).

The primary goals of CDP are to improve lymph circulation and prevent lymphatic stasis. CDP reduces swelling, heaviness, tightness, and pain, while increasing the range of motion (3). This approach has been shown to enhance sleep and QoL in individuals with BCRL (12, 14). In a study evaluating sleep and QoL before and after CDP in women with BCRL, significant improvements were observed in lymphedema stages, as well as sleep and QoL scores post-treatment (15).

Although many studies have examined sleep and QoL in women with BCRL, very few have focused on these outcomes following CDP. Existing studies often include all BCRL stages without comparing outcomes across different stages. CDP may have varying effects on sleep and QoL depending on the stage of BCRL, highlighting the need to investigate these effects in specific populations. Additionally, studies on the impact of CDP on sleep and QoL often lack follow-up data, leaving the Maintenance Phase unexplored.

This study aims to investigate the effects of CDP, including both the Decongestion and Maintenance phases, on sleep quality and QoL in women with Stage II BCRL.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged between 18 or 85 years,
* with a diagnosis of unilateral lymphedema in the upper extremity following breast cancer surgery
* stage 2 lymphedema confirmed by a doctor
* voluntary consent to participate in the study.

Exclusion Criteria:

* refusal to participate in the study
* development of lymphedema due to primary causes, presence of bilateral upper extremity lymphedema
* active soft tissue infection in the lymphedematous arm
* mental or cognitive disorders
* inability to communicate or cooperate
* acute deep vein thrombosis, arterial insufficiency in the upper extremity, systemic diseases that could cause edema other than lymphedema (e.g., renal failure, liver failure, heart failure)
* use of sleep medications or antidepressants

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 31 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | Baseline, 4th week and 1 month follow-up
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 18 questions that assess sleep quality over the past four weeks. It has seven subcomponents, each scored from 0 to 3. The subcomponents include subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction (17). The total score ranges from 0 to 21, with higher scores indicating worse sleep quality. A total score above 5 indicates poor sleep quality. The Turkish validity and reliability of the PSQI was established by Ağargün et al. (18).

SECONDARY OUTCOMES:
Quality of Life | Baseline, 4th week, 1 month follow-up
  Patients' quality of life will be assessed using the Lymphedema Quality of Life Questionnaire (LYMQoL). The LYMQoL consists of 4 subcomponents (function, mood, appearance, and symptoms) and 21 questions. Each question is evaluated on a 4-point Likert scale, where "1" indicates no effect and "4" indicates a high level of effect. The last question of the questionnaire assesses overall quality of life using a numeric visual analog scale (19). The total score is calculated by summing the scores of all questions and dividing by the number of questions. The total score ranges from 1 to 4, with higher scores indicating worse quality of life. The Turkish validity and reliability of the LYMQoL was established by Bakar et al. (20).
Tissue Dielectric Constant | Baseline, 4th week, 1 month follow-up
  The tissue dielectric constant (TDC) will be measured using the Moisturemeter-D device. The measurement method for TDC uses a co-axial reflection technique at a frequency of 300 MHz, which allows for the non-invasive measurement of free and bound local tissue fluid at effective penetration depths ranging from 0.5 to 5.0 mm (21). Measurements will be taken at a depth of 2.5 mm while the patient is in a supine position. TDC measurements will be made bilaterally at six reference points: the dorsum of the hand, the upper palmar wrist joint, 5 cm below and 7 cm above the elbow joint (forearm volar and arm volar), 7 cm below and 7 cm above the olecranon (forearm dorsal and arm dorsal), with three repeated measurements at each point. The TDC ratio will be calculated by dividing the affected side's TDC by the unaffected side's TDC. A TDC ratio of 1.20 is considered the threshold value for diagnosing lymphedema (22).
Volumetric Measurement | Baseline, 4th week, 1 month follow-up
  The volume of the extremity will be determined using the water displacement method. The measurement container will be filled with tap water to the overflow point. The participant will be asked to slowly submerge their arm into the container while leaning forward, ensuring the rod of the container fits between the second and third fingers. To prevent water spillage, participants will be instructed to avoid sudden movements. The displaced water will be transferred to another container, and the amount of displaced water will be recorded in milliliters (mL). Measurements will be made bilaterally, and the containers will be disinfected after each measurement. Residual extremity volume will be calculated using the formula: [(Affected extremity volume - Unaffected extremity volume) / Unaffected extremity volume] x 100. The volumetric measurement is considered the gold standard method for volume calculation in lymphedema patients (23).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bolu Abant Izzet Baysal University, Bolu, Bolu
  - Bolu Abant Izzet Baysal University, Bolu Merkez, Bolu

IPD SHARING:
Plan to Share IPD: No
Due to the Personal Data Protection Law, the data will not be shared.

REFERENCES:
- [Background] Konishi T, Tanabe M, Michihata N, Matsui H, Nishioka K, Fushimi K, Seto Y, Yasunaga H. Risk factors for arm lymphedema following breast cancer surgery: a Japanese nationwide database study of 84,022 patients. Breast Cancer. 2023 Jan;30(1):36-45. doi: 10.1007/s12282-022-01395-5. Epub 2022 Aug 23. PMID 35997891
- [Background] Janavlekar MG, Verma CV, Mistry HM. Effect of Complete Decongestive Therapy on Lymphoedema, Sleep Quality and Quality of Life in Metastatic Breast Cancer Patient - A Case Study. Indian J Palliat Care. 2022 Oct-Dec;28(4):439-442. doi: 10.25259/IJPC_78_2022. Epub 2022 Aug 25. PMID 36447505
- [Background] Deltombe T, Jamart J, Recloux S, Legrand C, Vandenbroeck N, Theys S, Hanson P. Reliability and limits of agreement of circumferential, water displacement, and optoelectronic volumetry in the measurement of upper limb lymphedema. Lymphology. 2007 Mar;40(1):26-34. PMID 17539462
- [Background] Naoum GE, Roberts S, Brunelle CL, Shui AM, Salama L, Daniell K, Gillespie T, Bucci L, Smith BL, Ho AY, Taghian AG. Quantifying the Impact of Axillary Surgery and Nodal Irradiation on Breast Cancer-Related Lymphedema and Local Tumor Control: Long-Term Results From a Prospective Screening Trial. J Clin Oncol. 2020 Oct 10;38(29):3430-3438. doi: 10.1200/JCO.20.00459. Epub 2020 Jul 30. PMID 32730184
- [Background] Ahn HR, Jeong HE, Jeong C, Kang SY, Jung SH, Youn HJ, Kim JS. Incidence and risk factors of breast cancer-related lymphedema in Korea: a nationwide retrospective cohort study. Int J Surg. 2024 Jun 1;110(6):3518-3526. doi: 10.1097/JS9.0000000000001278. PMID 38477155
- [Background] Corum M, Basoglu C, Korkmaz MD, Yildirim MA, Ones K. Effectiveness of Combined Complex Decongestive Therapy and Resistance Exercises in the Treatment of Lymphedema Associated with Breast Cancer and the Effect of Pain on Treatment Response. Lymphat Res Biol. 2021 Aug;19(4):383-390. doi: 10.1089/lrb.2020.0099. Epub 2021 Jan 15. PMID 33449865
- [Background] Thompson B, Gaitatzis K, Janse de Jonge X, Blackwell R, Koelmeyer LA. Manual lymphatic drainage treatment for lymphedema: a systematic review of the literature. J Cancer Surviv. 2021 Apr;15(2):244-258. doi: 10.1007/s11764-020-00928-1. Epub 2020 Aug 15. PMID 32803533
- [Background] Kligman L, Wong RK, Johnston M, Laetsch NS. The treatment of lymphedema related to breast cancer: a systematic review and evidence summary. Support Care Cancer. 2004 Jun;12(6):421-31. doi: 10.1007/s00520-004-0627-0. Epub 2004 Apr 17. PMID 15095073
- [Background] Mayrovitz HN. Assessing local tissue edema in postmastectomy lymphedema. Lymphology. 2007 Jun;40(2):87-94. PMID 17853619
- [Background] Mayrovitz HN, Davey S, Shapiro E. Local tissue water assessed by tissue dielectric constant: anatomical site and depth dependence in women prior to breast cancer treatment-related surgery. Clin Physiol Funct Imaging. 2008 Sep;28(5):337-42. doi: 10.1111/j.1475-097X.2008.00814.x. Epub 2008 Jun 5. PMID 18540873
- [Background] Bakar Y, Tugral A, Ozdemir O, Duygu E, Uyeturk U. Translation and Validation of the Turkish Version of Lymphedema Quality of Life Tool (LYMQOL) in Patients with Breast Cancer Related Lymphedema. Eur J Breast Health. 2017 Jul 1;13(3):123-128. doi: 10.5152/ejbh.2017.3522. eCollection 2017 Jul. PMID 28894851
- [Background] Carpenter JS, Andrykowski MA. Psychometric evaluation of the Pittsburgh Sleep Quality Index. J Psychosom Res. 1998 Jul;45(1):5-13. doi: 10.1016/s0022-3999(97)00298-5. PMID 9720850
- [Background] Kavak SK, Kavak EE. Fatigue and sleep quality improvement through complete decongestive therapy in postmastectomy lymphedema: An investigative analysis. Support Care Cancer. 2024 May 29;32(6):392. doi: 10.1007/s00520-024-08590-4. PMID 38806742
- [Background] Tzani I, Tsichlaki M, Zerva E, Papathanasiou G, Dimakakos E. Physiotherapeutic rehabilitation of lymphedema: state-of-the-art. Lymphology. 2018;51(1):1-12. PMID 30248726
- [Background] Sahbaz-Pirincci C, Cihan E, Duzlu-Ozturk U, Borman P, Dalyan M. Comparing complex decongestive therapy in patients with lymphedema of different causes by measuring: extremity volume, quality of life, and functionality. Cir Cir. 2024;92(3):354-361. doi: 10.24875/CIRU.23000330. PMID 38862116
- [Background] Tamam N, Al-Mugren KS, Alrebdi HI, Sulieman A, Abdelbasset WK. Evaluating the Quality of Life and Sleep Quality in Saudi Women with Breast Cancer-Related Lymphedema: A Cross-Sectional Correlational Study. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211046192. doi: 10.1177/15347354211046192. PMID 34541909
- [Background] Mete Civelek G, Akinci MG, Dalyan M. Evaluation of Sleep Quality, Depression, and Quality of Life in Patients with Breast Cancer Related Lymphedema. Lymphat Res Biol. 2023 Jun;21(3):289-295. doi: 10.1089/lrb.2022.0031. Epub 2022 Sep 29. PMID 36178954
- [Background] Kayiran O, De La Cruz C, Tane K, Soran A. Lymphedema: From diagnosis to treatment. Turk J Surg. 2017 Jun 1;33(2):51-57. doi: 10.5152/turkjsurg.2017.3870. eCollection 2017. PMID 28740950
- [Background] Duygu-Yildiz E, Bakar Y, Hizal M. The effect of complex decongestive physiotherapy applied with different compression pressures on skin and subcutaneous tissue thickness in individuals with breast cancer-related lymphedema: a double-blinded randomized comparison trial. Support Care Cancer. 2023 Jun 7;31(7):383. doi: 10.1007/s00520-023-07843-y. PMID 37285046
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Executive Committee of the International Society of Lymphology. The Diagnosis and Treatment of Peripheral Lymphedema: 2023 Consensus Document of The International Society of Lymphology. Lymphology. 2023;56(4):133-151. PMID 39207406
- [Background] Sharifi N, Ahmad S. Breast cancer-related lymphedema: A critical review on recent progress. Surg Oncol. 2024 Oct;56:102124. doi: 10.1016/j.suronc.2024.102124. Epub 2024 Aug 23. PMID 39208532
- See also: breast cancer statistics — https://gco.iarc.fr/today/en